CLINICAL TRIAL: NCT00272025
Title: Six Week Double Blind, Randomized Trial of Escitalopram Add On for Treatment Resistant Bipolar Depression
Brief Title: Treatment Resistant Bipolar Depression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lundbeck withdrew committment - expiring patents and prolonged inactivity
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSIY-207-05
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Bipolar Depression
Keywords: Bipolar Depression; Escitalopram; Mood Stabilizer; Atypical Antipsychotic
MeSH Terms: conditions — Bipolar Disorder | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): There is a 50% chance of being randomized to Escitalopram in addition to current atypical antipsychotic (minimum dose risperidone 3mg, olanzapine 10mg or seroquel 400mg) or mood stabilizer (lithium, epival or lamotrigine)
  Interventions: Drug: Escitalopram
- 2 (Placebo Comparator): to be filled in
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Escitalopram — 10mg to 20mg tablet daily for 6 weeks
  Other Names: Cipralex
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
To determine if adding Escitalopram to current mood stabilizer (MS) or atypical antipsychotic (AA) will improve in rates similar to or better than adding a placebo (inactive pill)in resistant bipolar patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of Bipolar Disorder and currently be in depressive state, and not responded to mood stabilizer or atypical antipsychotic alone or combined with an antidepressant medication.

Exclusion Criteria:

* Pregnant or breastfeeding
* History of seizure disorder or other unstable medical condition
* Received Electroconvulsive Therapy or Transcranial Magnetic Stimulation in the last three months
* Experienced hallucinations or delusions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rates when Escitalopram vs. placeboes added to the current mood stabilizer or antipsychotic medication | 6 weeks

SECONDARY OUTCOMES:
To evaluate efficacy, safety and tolerability of added Escitalopram, to a mood stabilizer or atypical antipsychotic. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roumen V. Milev, MD, Principal Investigator — Queen's University
Locations (1):
- Providence Care, Mental Health Services, Kingston, Ontario, Canada